CLINICAL TRIAL: NCT01196273
Title: HIV-HEART STUDY: A Prospective, Epidemiologic and Multicentre Trial to Determine the Cardiovascular Risk in HIV-infected Patients
Brief Title: Cardiovascular Diseases in HIV-infected Patients HIV-HEART Study: 5 Years Follow-up
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Collaborators: HIV-HEART Study Investigative Group (Unknown); German Heart Failure Network (Other); German Competence Network for HIV/AIDS (Other); German Federal Ministry of Education and Research (Other Government); Bristol-Myers Squibb (Industry); ViiV Healthcare (Industry); GlaxoSmithKline (Industry); Abbott (Industry); Boehringer Ingelheim (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: PD Dr. med. Till Neumann MD, Dr. med. Stefan Esser MD, University Hospital
Other Study IDs: 09-4085
Record Dates: First submitted 2010-05-07; First posted 2010-09-08 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2010-09

CONDITIONS: Coronary Heart Disease; Heart Failure; HIV; AIDS; Metabolic Syndrome
Keywords: Cardiac Diseases,; HIV-Infection,; AIDS,; Antiretroviral Therapy,; Cardiovascular Medication,; Risk Factors,; coronary heart disease,; heart failure,; metabolic syndrome
MeSH Terms: conditions — Coronary Disease; Heart Failure; Acquired Immunodeficiency Syndrome; Metabolic Syndrome; Heart Diseases | interventions — Restraint, Physical; Blood Specimen Collection; Health Care Economics and Organizations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stored blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Regional Ruhrgebiets Cohort
  Interventions: Other: Comprehensive non invasive cardiovascular examination

INTERVENTIONS:
Other: Comprehensive non invasive cardiovascular examination — The examination includes:
  * Anamnesis incl. admission form
  * Physical examination
  * Documentation of the medical therapy (incl. HAART)
  * Electrocardiogram
  * Transthoracic echocardiography
  * Exercise electrocardiogram
  * 6 minute walk test
  * Blood collection
  * Questionnaire to quality of life and health economics
  Other Names: The examination includes:; - Anamnesis incl. admission form; Physical examination; Documentation of the medical therapy (incl. HAART); Electrocardiogram; Transthoracic echocardiography; Exercise electrocardiogram; 6 minute walk test; Blood collection; Questionnaire to quality of life and health economics

SUMMARY:
HIV-infection is associated not only with a reduced function of the immune system, but also linked with diseases of other organ systems, in particular with the heart.

Heart conditions that have been described with HIV include

* Pericarditis,
* Pleural effusion
* Pulmonary hypertension (Venedic classification typ II)
* Dilated cardiomyopathy
* Heart failure
* Myocarditis
* Bacterial endocarditis
* Heart valve disorders In addition to previously stated disorders of the heart, the premature atherosclerosis of coronary arteries, a further even more important disease of the heart in this patient population, went into the focus of most HIV-researchers and physicians.

Premature atherosclerosis of coronary arteries results in coronary calcification, angina pectoris, myocardial infarction and sudden death. HIV-positive patients are at greater risk for a variety of heart-related conditions, including coronary artery disease. It is assumed, that HIV infection doubles the risk of a heart attack, according to recent research.

The reason for this link between HIV and heart-related conditions is unknown, but secondary infections that affect the heart muscle and coronary arteries have a greater chance of occurring in people with compromised immune systems. In addition, the HI-virus itself had been detected in the myocardium and might have an impact on the premature of cardiovascular diseases.

Furthermore, some of the medications used to treat HIV patients (antiretroviral therapy, ART) are assumed to have heart-related side effects.

Therefore, current treatment regimens for HIV infection have to be balanced against the marked benefits of antiretroviral treatment. Nevertheless, prevention of coronary heart disease should be integrated into current treatment procedures of HIV-infected patients.

The link between the heart and HIV is well established but not well understood. Therefore, further results are needed for efficient guidelines for the prevention, diagnostic and therapy of HIV-associated cardiovascular diseases.

DETAILED DESCRIPTION:
A comprehensive detailed description of the study procedures had been previously published (European Journal of medical research 2007;12:243-248).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Known HIV-infection
* Written informed consent

Exclusion Criteria:

* Acute cardiovascular disease
* Unstable hemodynamic status in the three weeks before inclusion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included outpatients who were at least 18 years of age, had a known HIV-infection and exhibited a stable disease status within 4 weeks before inclusion of the trial. Written informed consent was obtained from all participants.
Sampling Method: Non-Probability Sample
Enrollment: 1424 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Diseases in HIV-infected Patients | Baseline up to 5 years follow-up
  The detection of prevalence, aetiology, progression and severity of cardiovascular diseases - especially of coronary artery disease - in HIV-infected patients.

SECONDARY OUTCOMES:
Cardiovascular Disorders in HIV-infected Patients HIV-HEART | Baseline up to 5 years follow-up
  The study also investigates the impact of established risk factors and new HIV-specific risk factors of coronary artery disease such as, age, gender, virus-load, CD4-cell count. The HIV-HEART study will focus on the impact of medication including cardiovascular medication and antiretroviral medication. Further secondary objectives will be examined, including economic costs and quality of life of subjects with and without cardiovascular diseases in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Esser, MD, Principal Investigator — University Hospital, Essen; Till Neumann, MD, Principal Investigator — University Hospital, Essen
Locations (5):
- Germany (5):
  - University Hospital of Bochum, Department of Dermatology, Bochum
  - HIV Outpatient Department, Dortmund
  - University Hospital, Department of Dermatology and Venerology, Essen
  - University Hospital, West German Heart Center Essen, Essen
  - Clinical Coordinating Center Leipzig, Leipzig

REFERENCES:
- [Result] Neumann T. [HIV, AIDS and the cardiovascular risk]. Internist (Berl). 2008 Apr;49(4):429-30, 432-5. doi: 10.1007/s00108-008-2049-4. German. PMID 18305915
- [Result] Reinsch N, Buhr C, Krings P, Kaelsch H, Kahlert P, Konorza T, Neumann T, Erbel R; Competence Network of Heart Failure. Effect of gender and highly active antiretroviral therapy on HIV-related pulmonary arterial hypertension: results of the HIV-HEART Study. HIV Med. 2008 Aug;9(7):550-6. doi: 10.1111/j.1468-1293.2008.00602.x. Epub 2008 Jun 28. PMID 18557952
- [Result] Reinsch N, Buhr C, Krings P, Kaelsch H, Neuhaus K, Wieneke H, Erbel R, Neumann T; German Heart Failure Network. Prevalence and risk factors of prolonged QTc interval in HIV-infected patients: results of the HIV-HEART study. HIV Clin Trials. 2009 Jul-Aug;10(4):261-8. doi: 10.1310/hct1004-261. PMID 19723613
- [Result] Neumann T, Reinsch N, Neuhaus K, Brockmeyer N, Potthoff A, Esser S, Hower M, Neumann A, Mostardt S, Gelbrich G, Erbel R; fur die HIV-HEART-Studie sowie die Kompetenznetze Herzinsuffizienz und HIV/AIDS. [BNP in HIV-infected patients]. Herz. 2009 Dec;34(8):634-40. doi: 10.1007/s00059-009-3313-7. German. PMID 20024643
- [Result] Neumann T, Esser S, Potthoff A, Pankuweit S, Neumann A, Breuckmann F, Neuhaus K, Kondratieva J, Buck T, Muller-Tasch T, Wachter R, Prettin C, Gelbrich G, Herzog W, Pieske B, Rauchhaus M, Loffler M, Maisch B, Mugge A, Wasem J, Gerken G, Brockmeyer NH, Erbel R; HIV-HEART Study Investigative Group. Prevalence and natural history of heart failure in outpatient HIV-infected subjects: rationale and design of the HIV-HEART study. Eur J Med Res. 2007 Jun 27;12(6):243-8. PMID 17666313
- [Result] Breuckmann F, Neumann T, Kondratieva J, Wieneke H, Ross B, Nassenstein K, Barkhausen J, Kreuter A, Brockmeyer N, Erbel R. Dilated cardiomyopathy in two adult human immunodeficiency positive (HIV+) patients possibly related to highly active antiretroviral therapy (HAART). Eur J Med Res. 2005 Sep 12;10(9):395-9. PMID 16183552